CLINICAL TRIAL: NCT02763566
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Compare NSAI (Anastrozole or Letrozole) Plus Abemaciclib, a CDK4 and CDK6 Inhibitor, or Plus Placebo, and to Compare Fulvestrant Plus Abemaciclib or Plus Placebo in Postmenopausal Women With Hormone Receptor-Positive, HER2-Negative Locoregionally Recurrent or Metastatic Breast Cancer
Brief Title: A Study of Abemaciclib (LY2835219) in Participants With Breast Cancer
Acronym: MONARCH plus
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15530; I3Y-CR-JPBQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-05-04; First posted 2016-05-05 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Hormone Receptor-Positive; HER2-Negative; CDK4; CDK6
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Anastrozole; Letrozole; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) (Experimental): Abemaciclib given orally every 12 hours (Q12H) plus anastrozole or letrozole given orally every 24 hours (Q24H) on days 1 to 28 of a 28 day cycle. Participants receiving benefit may continue until disease progression.
  Interventions: Drug: Abemaciclib; Drug: Anastrozole; Drug: Letrozole
- Placebo + NSAI (Experimental): Placebo given orally Q12H plus anastrozole or letrozole given orally Q24H on days 1 to 28 of a 28 day cycle. Participants receiving benefit may continue until disease progression.
  Interventions: Drug: Anastrozole; Drug: Letrozole; Drug: Placebo
- Abemaciclib + Fulvestrant (Experimental): Abemaciclib given orally Q12H on days 1 to 28 of a 28 day cycle plus fulvestrant intramuscularly (IM) on days 1 and 15 of cycle 1, then on day 1 of cycle 2 and beyond. Participants receiving benefit may continue until disease progression.
  Interventions: Drug: Abemaciclib; Drug: Fulvestrant
- Placebo + Fulvestrant (Experimental): Placebo given orally Q12H on days 1 to 28 of a 28 day cycle plus fulvestrant IM on days 1 and 15 of cycle 1, then on day 1 of cycle 2 and beyond. Participants receiving benefit may continue until disease progression.
  Interventions: Drug: Placebo; Drug: Fulvestrant

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: Abemaciclib + Fulvestrant; Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI)
Drug: Anastrozole — Administered orally
  Arms: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI); Placebo + NSAI
Drug: Letrozole — Administered orally
  Arms: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI); Placebo + NSAI
Drug: Placebo — Administered orally
  Arms: Placebo + Fulvestrant; Placebo + NSAI
Drug: Fulvestrant — Administered intramuscularly
  Arms: Abemaciclib + Fulvestrant; Placebo + Fulvestrant

SUMMARY:
The main purpose of this study is to evaluate the efficacy of the study drug abemaciclib in postmenopausal women with hormone receptor-positive (HR+), human epidermal growth factor receptor 2-negative (HER2-) locoregionally recurrent or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of HR+, HER2- breast cancer. Although not required as a protocol procedure, metastatic disease should be considered for biopsy whenever possible to reassess hormone receptor (HR) and human epidermal growth factor receptor 2 (HER2) status if clinically indicated.

  * To fulfill the requirement for HR+ disease, a breast cancer must express, by immunohistochemistry (IHC), at least 1 of the HRs (estrogen receptor [ER], progesterone receptor [PgR]) as defined in the relevant American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines.
  * To fulfill the requirement of HER2- disease, a breast cancer must not demonstrate, at initial diagnosis or upon subsequent biopsy, overexpression of HER2 by either IHC or in-situ hybridization as defined in the relevant ASCO/CAP guidelines.
* Meet either Inclusion Criterion (2a) or Inclusion Criterion (2b). Participants meeting Inclusion Criterion 2a will be enrolled in Cohort A and participants meeting Inclusion Criterion 2b will be enrolled in Cohort B.
* (2a) Have locoregionally recurrent disease not amenable to resection or radiation therapy with curative intent or metastatic disease.

  * Relapsed with radiologic evidence of progression more than 1 year from completion of adjuvant endocrine therapy and have received no prior endocrine therapy for locoregionally recurrent or metastatic disease (Note: prior adjuvant endocrine therapy for localized disease may have included, but is not limited to, anti-estrogens or aromatase inhibitors. In addition, a participant may be enrolled if she has received ≤2 weeks of NSAI in this disease setting immediately preceding screening and agrees to discontinue NSAI until study treatment initiation.) OR
  * Presented with de novo metastatic breast cancer (mBC) and not received any prior endocrine therapy. OR
* Relapsed with radiologic evidence of progression less than 1 year from completion of or while receiving adjuvant endocrine therapy (except for letrozole or anastrozole) and have received no prior endocrine therapy for locoregionally recurrent or metastatic disease.
* (2b) Have locoregionally recurrent disease not amenable to resection or radiation therapy with curative intent or metastatic disease.

  * Relapsed with radiologic evidence of progression while receiving neoadjuvant or adjuvant endocrine therapy, with no subsequent endocrine therapy received following progression OR
  * Relapsed with radiologic evidence of progression within 1 year from completion of adjuvant endocrine therapy, with no subsequent endocrine therapy received following progression OR
  * Relapsed with radiologic evidence of progression more than 1 year from completion of adjuvant endocrine therapy and then subsequently relapsed with radiologic evidence of progression after receiving treatment with either an antiestrogen or an aromatase inhibitor as firstline endocrine therapy for metastatic disease. Participants may not have received more than 1 line of endocrine therapy or any prior chemotherapy for metastatic disease OR
  * Presented with de novo metastatic disease and then relapsed with radiologic evidence of progression after receiving treatment with either an antiestrogen or an aromatase inhibitor as first-line endocrine therapy for metastatic disease. Participants may not have received more than 1 line of endocrine therapy or any prior chemotherapy for metastatic disease.
* Have postmenopausal status defined as meeting at least 1 of the following:

  * Prior bilateral oophorectomy
  * Age ≥60 years
  * Age <60 years and amenorrheic for at least 12 months (in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression) and follicle-stimulating hormone (FSH) and estradiol levels in the postmenopausal range.
* Have 1 of the following, as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1:

  * Measurable disease
  * Nonmeasurable bone-only disease. Nonmeasurable bone-only disease may include any of the following: blastic bone lesions, lytic bone lesions without a measurable soft tissue component, or mixed lytic-blastic bone lesions without a measurable soft tissue component.
* Have a performance status (PS) of ≤1 on the Eastern Cooperative Oncology (ECOG) scale.
* Have adequate organ function, including:

  * Hematologic: absolute neutrophil count (ANC) ≥1.5 × 109/Liter (L), platelets

    ≥100 × 109/L, and hemoglobin ≥8 g/deciliter (dL). Participants may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator; however, initial study drug treatment must not begin earlier than the day after the erythrocyte transfusion.
  * Hepatic: Total bilirubin ≤1.5 times the upper limit of normal (ULN) and alanine aminotransferase (ALT) and aspartate aminotransferase (AST)

    ≤3.0 times ULN (or ALT and AST ≤5 times ULN if liver metastases are present).
  * Renal: serum creatinine ≤1.5 times ULN.
* Have discontinued previous localized radiotherapy for palliative purposes or for lytic lesions at risk of fracture at least 2 weeks prior to randomization and recovered from the acute effects of therapy (until the toxicity resolves to either baseline or at least Grade 1) except for residual alopecia or peripheral neuropathy.
* Are able to swallow capsules.
* Are reliable, willing to be available for the duration of the study, and willing to follow study procedures.

Exclusion Criteria:

* Have visceral crisis, lymphangitic spread, or leptomeningeal carcinomatosis. Visceral crisis is not the mere presence of visceral metastases, but implies severe organ dysfunction as assessed by symptoms and signs, laboratory studies, and rapid progression of the disease.
* Have inflammatory breast cancer.
* Have clinical evidence or a history of central nervous system (CNS) metastasis. Screening test is not required for enrollment.
* Are currently receiving or have previously received chemotherapy for locoregionally recurrent or metastatic breast cancer. (Note: Participants may be enrolled if they received prior [neo]adjuvant chemotherapy for localized disease.)
* Have received prior treatment with everolimus or fulvestrant (for Cohort B only).
* Have received prior treatment with any cyclin-dependent kinases 4 and 6 (CDK4 and CDK6) inhibitor (or participated in any CDK4 and CDK6 inhibitor clinical trial for which treatment assignment is still blinded).
* Have initiated bisphosphonates or approved Receptor activator of nuclear factor kappa-B ligand (RANK-L) targeted agents <7 days prior to randomization.
* Are currently enrolled in a clinical trial involving an investigational product (IP) or non-approved use of a drug or device (other than the IP/device used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study. If a participant is currently enrolled in a clinical trial involving non-approved use of a device, then agreement with the investigator and Eli Lilly and Company (Lilly) clinical research physician (CRP) is required to establish eligibility.
* Have received treatment with a drug that has not received regulatory approval for any indication within 14 or 21 days of randomization for a nonmyelosuppressive or myelosuppressive agent, respectively.
* Have had major surgery within 14 days prior to randomization to allow for post-operative healing of the surgical wound and site(s).
* Have received recent (within 28 days prior to randomization) live attenuated vaccines such as yellow fever vaccine.
* Have serious preexisting medical conditions that, in the judgment of the investigator, would preclude participation in this study (eg, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis).
* Have a personal history within the last 12 months of any of the following conditions: syncope of cardiovascular etiology, ventricular tachycardia, ventricular fibrillation, or sudden cardiac arrest.
* Have a history of any other cancer (except nonmelanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission with no therapy for a minimum of 3 years.
* Have received an autologous or allogeneic stem-cell transplant.
* Have clinical evidence of active bacterial or fungal infection or active viral infection that, in the judgment of the investigator, would preclude participation in this study (eg, human immunodeficiency virus [HIV] or viral hepatitis). Screening test is not required for enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2028-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (45):
- Brazil (6):
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia, Ijuí, Rio Grande do Sul
  - Centro Gaucho Integrado De Oncologia, Hematologia, Ensino E Pesquisa, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
  - Clínica de Pesquisa e Centro de Estudos em Ginecologia Oncológica e Mamária LTDA, São Paulo
- China (28):
  - Afflilated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Provincial Cancer hospital, Fuzhou, Fujian
  - Fuzhou General hospital of Nanjing Military Command, Fuzhou, Fujian
  - Guangdong Province People's Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Caner Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Wuhan Union Hospital Cancer Center, Wuhan, Hubei
  - Tongji Hospital Tongji Medical, Science & Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jilin Province Tumor Hospital, Changchun, Jilin
  - The 2nd Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital&Institute, Shenyang, Liaoning
  - The first affiliated hospital of China medical university, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The Second Affiliate Hospital of Zhejiang University School of medicine, Hangzhou, Zhejiang
- India (8):
  - The Gujarat Cancer & Research Institute (GCRI), Ahmedabad, Gujarat
  - Healthcare Global Enterprises Limited (HCG), Bangalore, Karnataka
  - M S Ramaiah Medical College Hospitals, Bangalore, Karnataka
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Jehangir Hospital, Pune, Maharashtra
  - Dr. B. L. Kapur Memorial Hospital, New Delhi, National Capital Territory of Delhi
  - Christian Medical College Vellore, Ranipet, Tamil Nadu
  - Medica Superspecialty Hospital, Kolkata, West Bengal
- South Africa (3):
  - The Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Eastleigh Breast Care Center, Pretoria, Gauteng
  - Sandton Oncology Centre, Johannesburg

REFERENCES:
- [Derived] Hu X, Zhang Q, Sun T, Yin Y, Li H, Yan M, Tong Z, Li M, Teng Y, Oppermann CP, Kanakasetty GB, Portugal MC, Yang L, Zhang W, Jiang Z. Abemaciclib plus non-steroidal aromatase inhibitor or fulvestrant in women with HR+/HER2- advanced breast cancer: Final results of the randomized phase III MONARCH plus trial. Chin Med J (Engl). 2025 Jun 20;138(12):1477-1486. doi: 10.1097/CM9.0000000000003151. Epub 2024 Oct 10. PMID 39385327
- [Derived] Zhang QY, Sun T, Yin YM, Li HP, Yan M, Tong ZS, Oppermann CP, Liu YP, Costa R, Li M, Cheng Y, Ouyang QC, Chen X, Liao N, Wu XH, Wang XJ, Feng JF, Hegg R, Kanakasetty GB, Coccia-Portugal MA, Han RB, Lu Y, Chi HD, Jiang ZF, Hu XC. MONARCH plus: abemaciclib plus endocrine therapy in women with HR+/HER2- advanced breast cancer: the multinational randomized phase III study. Ther Adv Med Oncol. 2020 Oct 22;12:1758835920963925. doi: 10.1177/1758835920963925. eCollection 2020. PMID 33149768
- See also: A Study of Abemaciclib (LY2835219) in Participants With Breast Cancer — https://trials.lillytrialguide.com/en-US/trial/5gZx1MGGogIqeyI6uuKOO

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who died due to any cause or disease progression or alive and on study at conclusion but off treatment are considered as completed.
Groups:
- Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI): Participants received Abemaciclib orally every 12 hours (Q12H) plus anastrozole or letrozole given orally every 24 hours (Q24H) on days 1 to 28 of a 28 day cycle.
- Placebo + NSAI: Participants received Placebo orally Q12H plus anastrozole or letrozole given orally Q24H on days 1 to 28 of a 28 day cycle.
- Abemaciclib + Fulvestrant: Participants received Abemaciclib orally Q12H on days 1 to 28 of a 28 day cycle plus fulvestrant intramuscularly (IM) on days 1 and 15 of cycle 1, then on day 1 of cycle 2 and beyond.
- Placebo + Fulvestrant: Participants received Placebo orally Q12H on days 1 to 28 of a 28 day cycle plus fulvestrant IM on days 1 and 15 of cycle 1, then on day 1 of cycle 2 and beyond.
Period: Overall Study
Arm/Group | Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) | Placebo + NSAI | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Started | 207 | 99 | 104 | 53
Completed | 89 | 60 | 50 | 39
Not Completed | 118 | 39 | 54 | 14
Not completed — Lost to Follow-up | 1 | 4 | 0 | 1
Not completed — On study treatment at study conclusion | 114 | 34 | 54 | 13
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) | Placebo + NSAI | Abemaciclib + Fulvestrant | Placebo + Fulvestrant | Total
Number analyzed (Participants) | 207 | 99 | 104 | 53 | 463
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (10.8) | 55.5 (9.8) | 59.7 (8.5) | 58.2 (10.3) | 57.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 99 | 104 | 53 | 463
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 207 | 99 | 104 | 53 | 463
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 182 | 89 | 94 | 48 | 413
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 1 | 5
  White | 24 | 8 | 8 | 4 | 44
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 164 | 82 | 89 | 45 | 380
  Brazil | 21 | 8 | 10 | 5 | 44
  South Africa | 4 | 2 | 0 | 1 | 7
  India | 18 | 7 | 5 | 2 | 32

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) (Abemaciclib + NSAI & Placebo NSAI)
Description: Progression-free survival time was measured from randomization until the date of objective progression as defined by Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1), or death from any cause. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. Patients who have neither progressed nor died were censored at the day of their last radiographic tumor assessment, if available, or date of randomization if no post-baseline radiographic assessment is available.
Time Frame: Randomization to Measured Progressive Disease or Death (up to 26 Months)
Population: All randomized participants in Abemaciclib + NSAI & Placebo NSAI arms. Censored participants: 141 in Abemaciclib + NSAI, 46 in Placebo + NSAI.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) | Placebo + NSAI
Number analyzed (Participants) | 207 | 99
Months | NA [22.32 to NA] — Median and Upper bound were not estimable due to Immature data. | 14.73 [11.21 to 18.87]
Statistical Analysis 1: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Test type: Superiority; p = 0.0001, Log Rank; Hazard Ratio (HR) = 0.499, 95% CI 2-sided [0.346 to 0.719]

2. Secondary Outcome: Progression Free Survival (PFS) (Abemaciclib + Fulvestrant and Placebo + Fulvestrant Arms)
Description: as for outcome 1
Time Frame: Randomization to Measured Progressive Disease or Death (up to 26 Months)
Population: All randomized participants in Abemaciclib + Fulvestrant and Placebo + Fulvestrant arms.
  Censored participants: 58 in Abemaciclib + Fulvestrant, 17 in Placebo + Fulvestrant.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 104 | 53
Months | 11.47 [9.53 to NA] — Upper bound was not estimable due to Immature data. | 5.59 [3.65 to 7.69]
Statistical Analysis 1: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.376, 95% CI 2-sided [0.240 to 0.588]

3. Secondary Outcome: Overall Survival (OS)
Time Frame: Randomization to Date of Death from Any Cause (Estimated up to 38 Months)
Reporting Status: Not Posted

4. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)]
Description: Objective response rate is the percentage of participants with a BOR of CR or PR as defined by RECIST v1.1. CR is defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions.
Time Frame: Randomization to Measured Progressive Disease (up to 26 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) | Placebo + NSAI | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 207 | 99 | 104 | 53
percentage of participants | 56.0 [49.3 to 62.8] | 30.3 [21.3 to 39.4] | 38.5 [29.1 to 47.8] | 7.5 [0.4 to 14.7]
Statistical Analysis 1: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

5. Secondary Outcome: Duration of Response (DoR)
Time Frame: Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Estimated up to 38 Months)
Reporting Status: Not Posted

6. Secondary Outcome: Percentage of Participants Who Exhibit Stable Disease (SD) or CR or PR [Disease Control Rate (DCR)]
Description: Disease control rate (DCR) is the percentage of participants with a best overall response of CR, PR or SD as defined by RECIST v1.1. CR is defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Randomization to Measured Progressive Disease (up to 26 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) | Placebo + NSAI | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 207 | 99 | 104 | 53
percentage of participants | 91.3 [87.5 to 95.1] | 82.8 [75.4 to 90.3] | 92.3 [87.2 to 97.4] | 69.8 [57.5 to 82.2]
Statistical Analysis 1: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Test type: Superiority; p = 0.0456, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel

7. Secondary Outcome: Percentage of Participants With Best Overall Response of CR, PR, or SD With Duration of SD for at Least 6 Months [Clinical Benefit Rate (CBR)]
Description: Clinical benefit rate (CBR) is the percentage of participants with a BOR of CR or PR, or SD for at least 6 months. CR is defined as the disappearance of all target and non-target lesions & no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Randomization to Measured Progressive Disease (up to 26 Months)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) | Placebo + NSAI | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 207 | 99 | 104 | 53
percentage of participants | 82.6 [77.4 to 87.8] | 62.6 [53.1 to 72.2] | 77.9 [69.9 to 85.9] | 45.3 [31.9 to 58.7]
Statistical Analysis 1: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

8. Secondary Outcome: Change From Randomization in Symptom Burden on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30)
Description: consists of 30 items covered by 1 of 3 dimensions:
  1. Global health status/quality of life (2 items) with scores ranging from 1 (Very Poor) to 7 (Excellent).
  2. Functional scales (15 total items addressing either physical, role, emotional, cognitive, or social functioning), each item scores ranging from 1 (not at all) to 4 (very much)
  3. Symptom scales (13 total items addressing either fatigue, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, or financial impact), each item scores ranging from 1 (not at all) to 4 (very much).
  Raw scores are linearly converted to a 0-100 scale with higher scores reflecting higher levels of function/QOL or higher levels of symptom burden.
Time Frame: Baseline through 19 Months
Population: All randomized participants who received at least one dose of study drug and had baseline EORTC-QLQ-C30 measurement.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo + NSAI: Participants received Placebo orally Q12H plus anastrozole or letrozole given orally Q24H on days 1 to 28 of a 28 day cycle. Participants receiving benefit may continue until disease progression.
Arm/Group | Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) | Placebo + NSAI | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 202 | 97 | 97 | 51
score on a scale
  Global Health Status | 2.38 (0.99) | 4.26 (1.47) | -0.35 (1.41) | 3.12 (2.07)
  Functional Scales - Physical Functioning | -0.78 (0.82) | -0.01 (1.21) | -1.11 (1.06) | -2.70 (1.54)
  Functional Scales - Role Functioning | -1.69 (1.20) | -1.38 (1.79) | -3.76 (1.35) | -2.04 (1.95)
  Functional Scales - Emotional Functioning | 1.57 (0.98) | -0.10 (1.44) | 0.43 (1.27) | 0.18 (1.85)
  Functional Scales - Cognitive Functioning | -2.89 (0.90) | -0.72 (1.35) | -3.52 (1.35) | -1.10 (1.96)
  Functional Scales - Social Functioning | -2.45 (1.19) | -1.57 (1.75) | -2.03 (1.71) | -2.67 (2.44)
  Symptom Scales - Fatigue | 1.63 (0.95) | 0.06 (1.40) | 4.19 (1.44) | 1.46 (2.08)
  Symptom Scales - Nausea and Vomiting | 0.62 (0.60) | -0.33 (0.88) | 4.26 (1.10) | 1.67 (1.65)
  Symptom Scales - Pain | -5.44 (0.91) | -4.90 (1.35) | -2.82 (1.36) | -0.17 (2.01)
  Symptom Scales - Dyspnoea | 2.51 (1.02) | 0.35 (1.53) | -1.66 (1.27) | 0.83 (1.92)
  Symptom Scales - Insomnia | -0.87 (1.07) | -0.05 (1.60) | 1.53 (1.59) | -0.44 (2.42)
  Symptom Scales - Appetite | 4.19 (0.97) | -1.47 (1.44) | 8.67 (1.63) | 1.21 (2.42)
  Symptom Scales - Constipation | -3.05 (0.98) | -1.49 (1.46) | -1.63 (1.31) | 0.65 (1.88)
  Symptom Scales - Diarrhoea | 15.72 (0.85) | -0.10 (1.27) | 16.03 (1.26) | -1.80 (1.95)
  Symptom Scales - Financial Difficulties | -3.02 (1.65) | -1.27 (2.46) | -6.36 (1.76) | -9.35 (2.59)
Statistical Analysis 1: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Global Health Status; Test type: Superiority; p = 0.287, Mixed Models Analysis; LSMean Difference = -1.89, 95% CI 2-sided [-5.36 to 1.59], Standard Error of Mean 1.77
Statistical Analysis 2: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Functional Scales - Physical functioning; Test type: Superiority; p = 0.597, Mixed Models Analysis; LSMean Difference = -0.77, 95% CI 2-sided [-3.64 to 2.10], Standard Error of Mean 1.46
Statistical Analysis 3: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Functional Scales - Role Functioning; Test type: Superiority; p = 0.885, Mixed Models Analysis; LSMean Difference = -0.31, 95% CI 2-sided [-4.55 to 3.93], Standard Error of Mean 2.15
Statistical Analysis 4: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Functional Scales - Emotional Functioning; Test type: Superiority; p = 0.340, Mixed Models Analysis; LSMean Difference = 1.67, 95% CI 2-sided [-1.77 to 5.10], Standard Error of Mean 1.74
Statistical Analysis 5: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Functional Scales - Cognitive Functioning; Test type: Superiority; p = 0.182, Mixed Models Analysis; LSMean Difference = -2.17, 95% CI 2-sided [-5.37 to 1.03], Standard Error of Mean 1.62
Statistical Analysis 6: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Test type: Superiority; p = 0.678, Mixed Models Analysis; LSMean Difference = -0.88, 95% CI 2-sided [-5.05 to 3.29], Standard Error of Mean 2.12
Statistical Analysis 7: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Symptom Scales - Fatigue; Test type: Superiority; p = 0.355, Mixed Models Analysis; LSMean Difference = 1.57, 95% CI 2-sided [-1.77 to 4.91], Standard Error of Mean 1.70
Statistical Analysis 8: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Symptom Scales - Nausea and Vomiting; Test type: Superiority; p = 0.372, Mixed Models Analysis; LSMean Difference = 0.95, 95% CI 2-sided [-1.14 to 3.03], Standard Error of Mean 1.06
Statistical Analysis 9: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Symptom Scales - Pain; Test type: Superiority; p = 0.740, Mixed Models Analysis; LSMean Difference = 0.740, 95% CI 2-sided [-3.75 to 2.66], Standard Error of Mean 1.63
Statistical Analysis 10: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Symptom Scales - Dyspnoea; Test type: Superiority; p = 0.240, Mixed Models Analysis; LSMean Difference = 2.16, 95% CI 2-sided [-1.46 to 5.78], Standard Error of Mean 1.84
Statistical Analysis 11: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Symptom scales - Insomnia; Test type: Superiority; p = 0.673, Mixed Models Analysis; LSMean Difference = -0.81, 95% CI 2-sided [-4.60 to 2.97], Standard Error of Mean 1.92
Statistical Analysis 12: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Symptom Scales - Appetite; Test type: Superiority; p = 0.001, Mixed Models Analysis; LSMean Difference = 5.65, 95% CI 2-sided [2.23 to 9.07], Standard Error of Mean 1.74
Statistical Analysis 13: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Symptom Scales - Constipation; Test type: Superiority; p = 0.375, Mixed Models Analysis; LSMean Difference = -1.57, 95% CI 2-sided [-5.04 to 1.91], Standard Error of Mean 1.76
Statistical Analysis 14: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Symptom Scales - Diarrhoea; Test type: Superiority; p = 0.000, Mixed Models Analysis; LSMean Difference = 15.82, 95% CI 2-sided [12.81 to 18.84], Standard Error of Mean 1.53
Statistical Analysis 15: Comparison: Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) vs Placebo + NSAI; Symptom Scales - Financial Difficulties; Test type: Superiority; p = 0.557, Mixed Models Analysis; LSMean Difference = -1.75, 95% CI 2-sided [-7.59 to 4.10], Standard Error of Mean 2.97
Statistical Analysis 16: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Global Health Status; Test type: Superiority; p = 0.169, Mixed Models Analysis; LSMean Difference = -3.47, 95% CI 2-sided [-8.43 to 1.49], Standard Error of Mean 2.51
Statistical Analysis 17: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Functional Scales - Physical Functioning; Test type: Superiority; p = 0.400, Mixed Models Analysis; LSMean Difference = 1.58, 95% CI 2-sided [-2.12 to 5.29], Standard Error of Mean 1.87
Statistical Analysis 18: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Functional Scales - Role functioning; Test type: Superiority; p = 0.472, Mixed Models Analysis; LSMean Difference = -1.72, 95% CI 2-sided [-6.42 to 2.99], Standard Error of Mean 2.38
Statistical Analysis 19: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Functional Scales - Emotional Functioning; Test type: Superiority; p = 0.310, Mixed Models Analysis; LSMean Difference = -2.42, 95% CI 2-sided [-7.12 to 2.28], Standard Error of Mean 0.310
Statistical Analysis 20: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Functional Scales - Social Functioning; Test type: Superiority; p = 0.830, Mixed Models Analysis; LSMean Difference = 0.64, 95% CI 2-sided [-5.26 to 6.55], Standard Error of Mean 2.98
Statistical Analysis 21: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Symptom Scales - Fatigue; Test type: Superiority; p = 0.281, Mixed Models Analysis; LSMean Difference = 2.73, 95% CI 2-sided [-2.26 to 7.72], Standard Error of Mean 2.52
Statistical Analysis 22: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Symptom Scales - Nausea and Vomiting; Test type: Superiority; p = 0.194, Mixed Models Analysis; LSMean Difference = 2.59, 95% CI 2-sided [-1.33 to 6.52], Standard Error of Mean 1.99
Statistical Analysis 23: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Symptom Scales - Pain; Test type: Superiority; p = 0.275, Mixed Models Analysis; LSMean Difference = -2.66, 95% CI 2-sided [-7.45 to 2.14], Standard Error of Mean 2.42
Statistical Analysis 24: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Symptom Scales - Dyspnoea; Test type: Superiority; p = 0.280, Mixed Models Analysis; LSMean Difference = -2.49, 95% CI 2-sided [-7.04 to 2.06], Standard Error of Mean 4.39
Statistical Analysis 25: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Symptom Scales - Insomnia; Test type: Superiority; p = 0.499, Mixed Models Analysis; LSMean Difference = 1.97, 95% CI 2-sided [-3.78 to 7.72], Standard Error of Mean 2.90
Statistical Analysis 26: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Symptom Scales - Appetite; Test type: Superiority; p = 0.012, Mixed Models Analysis; LSMean Difference = 7.46, 95% CI 2-sided [1.68 to 13.23], Standard Error of Mean 2.92
Statistical Analysis 27: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Symptom Scales - Constipation; Test type: Superiority; p = 0.321, Mixed Models Analysis; LSMean Difference = -2.28, 95% CI 2-sided [-6.83 to 2.27], Standard Error of Mean 2.29
Statistical Analysis 28: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Symptom Scales - Diarrhoea; Test type: Superiority; p = 0.000, Mixed Models Analysis; LSMean Difference = 17.83, 95% CI 2-sided [13.25 to 22.41], Standard Error of Mean 2.32
Statistical Analysis 29: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Symptom Scales - Financial DIfficulties; Test type: Superiority; p = 0.342, Mixed Models Analysis; LSMean Difference = 2.99, 95% CI 2-sided [-3.21 to 9.19], Standard Error of Mean 3.14
Statistical Analysis 30: Comparison: Abemaciclib + Fulvestrant vs Placebo + Fulvestrant; Functional Scales - Cognitive functioning; Test type: Superiority; p = 0.310, Mixed Models Analysis; LSMean Difference = -2.42, 95% CI 2-sided [-7.12 to 2.28], Standard Error of Mean 2.38

9. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve of Abemaciclib, Its Metabolites (M2 & M20)
Description: Pharmacokinetics (PK): Area Under the Concentration Curve of Abemaciclib and its Metabolites LSN2839567 (M2) & LSN3106726 (M20) was reported.
  C=Cycle, D=day;
Time Frame: C1D1 post dose, C2D1 post dose, C3D1 predose, C4D1 predose
Population: All randomized participants who received at least one dose of Abemaciclib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per Millilitre (ng*h/mL)
Arm/Group | Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) | Abemaciclib + Fulvestrant
Number analyzed (Participants) | 204 | 101
Nanogram*hour per Millilitre (ng*h/mL)
  Abemaciclib | 2720 (40) | 2740 (57)
  LSN2839567 (M2) | 1080 (84) | 861 (120)
  LSN3106726 (M20) | 1970 (81) | 1570 (110)

ADVERSE EVENTS:
Time Frame: Up to 28 Months
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) | Placebo + NSAI | Abemaciclib + Fulvestrant | Placebo + Fulvestrant
All-Cause Mortality (participants affected / at risk) | 20/205 | 10/99 | 8/104 | 9/53
Serious Adverse Events (participants affected / at risk) | 40/205 | 9/99 | 16/104 | 4/53
Other Adverse Events (participants affected / at risk) | 204/205 | 85/99 | 103/104 | 39/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) (N=205) | Placebo + NSAI (N=99) | Abemaciclib + Fulvestrant (N=104) | Placebo + Fulvestrant (N=53)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 6 (10) | 1 (1) | 2 (3) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urostomy complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iiird nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib + Nonsteroidal Aromatase Inhibitor (NSAI) (N=205) | Placebo + NSAI (N=99) | Abemaciclib + Fulvestrant (N=104) | Placebo + Fulvestrant (N=53)
Anaemia (Blood and lymphatic system disorders) | 127 (462) | 20 (39) | 73 (206) | 8 (14)
Lacrimation increased (Eye disorders) | 10 (13) | 0 (0) | 6 (7) | 0 (0)
Vision blurred (Eye disorders) | 13 (13) | 3 (10) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 36 (101) | 9 (21) | 15 (32) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 24 (35) | 0 (0) | 6 (10) | 0 (0)
Constipation (Gastrointestinal disorders) | 21 (31) | 8 (11) | 5 (12) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 164 (960) | 15 (45) | 82 (449) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 11 (12) | 3 (4) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 54 (75) | 19 (30) | 19 (25) | 9 (17)
Stomatitis (Gastrointestinal disorders) | 21 (44) | 2 (2) | 12 (18) | 1 (1)
Toothache (Gastrointestinal disorders) | 7 (11) | 5 (5) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 29 (38) | 13 (19) | 20 (29) | 5 (6)
Fatigue (General disorders) | 60 (87) | 25 (41) | 24 (35) | 8 (11)
Influenza like illness (General disorders) | 30 (42) | 13 (18) | 12 (13) | 2 (6)
Localised oedema (General disorders) | 7 (9) | 0 (0) | 10 (14) | 2 (2)
Malaise (General disorders) | 19 (38) | 7 (11) | 9 (11) | 3 (4)
Oedema peripheral (General disorders) | 20 (28) | 2 (2) | 3 (4) | 2 (2)
Pain (General disorders) | 21 (26) | 7 (10) | 6 (8) | 8 (14)
Pyrexia (General disorders) | 19 (25) | 11 (13) | 9 (15) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 31 (39) | 22 (31) | 14 (17) | 4 (4)
Alanine aminotransferase increased (Investigations) | 71 (143) | 23 (40) | 36 (68) | 12 (17)
Aspartate aminotransferase increased (Investigations) | 71 (142) | 21 (35) | 32 (53) | 14 (19)
Blood alkaline phosphatase increased (Investigations) | 24 (39) | 12 (17) | 6 (7) | 4 (5)
Blood cholesterol increased (Investigations) | 12 (23) | 1 (1) | 7 (9) | 1 (1)
Blood creatinine increased (Investigations) | 24 (52) | 2 (7) | 22 (38) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 11 (18) | 5 (6) | 5 (14) | 4 (4)
Lymphocyte count decreased (Investigations) | 34 (91) | 4 (7) | 22 (56) | 1 (3)
Monocyte count decreased (Investigations) | 11 (29) | 1 (3) | 8 (17) | 0 (0)
Neutrophil count decreased (Investigations) | 164 (953) | 20 (44) | 84 (392) | 10 (29)
Platelet count decreased (Investigations) | 90 (247) | 7 (15) | 43 (100) | 5 (13)
Weight decreased (Investigations) | 38 (64) | 4 (5) | 15 (22) | 1 (2)
Weight increased (Investigations) | 14 (28) | 9 (15) | 3 (3) | 2 (2)
White blood cell count decreased (Investigations) | 156 (891) | 27 (58) | 86 (374) | 12 (24)
Decreased appetite (Metabolism and nutrition disorders) | 48 (70) | 11 (18) | 23 (34) | 6 (8)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 8 (18) | 3 (3) | 8 (9) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 (12) | 5 (5) | 4 (6) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 11 (18) | 2 (6) | 4 (5) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 25 (56) | 4 (5) | 9 (18) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (21) | 13 (19) | 7 (10) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (18) | 9 (10) | 5 (5) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (11) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (13) | 5 (7) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (16) | 7 (8) | 3 (3) | 5 (11)
Dizziness (Nervous system disorders) | 17 (22) | 8 (15) | 5 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 14 (16) | 2 (3) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 22 (27) | 13 (23) | 6 (7) | 5 (9)
Insomnia (Psychiatric disorders) | 25 (40) | 18 (20) | 13 (16) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 5 (7) | 6 (11) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (41) | 9 (11) | 12 (14) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (27) | 4 (4) | 2 (3) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 2 (2) | 1 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 17 (19) | 5 (6) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 24 (36) | 5 (6) | 9 (9) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 19 (24) | 0 (0) | 4 (4) | 0 (0)
Hot flush (Vascular disorders) | 11 (13) | 8 (8) | 3 (4) | 1 (1)
Hypertension (Vascular disorders) | 14 (27) | 9 (12) | 4 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT02763566/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT02763566/SAP_001.pdf